CLINICAL TRIAL: NCT03428139
Title: Role of Alpha Lipoic Acid Combined With Pulsed Radiofrequency in Treatment of Chronic Lumbosacral Radicular Pain: Prospective, Randomized Study
Brief Title: Alpha Lipoic Acid and Chronic Lumbosacral Radicular Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0000871245
Record Dates: First submitted 2018-01-27; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Radicular; Neuropathic, Lumbar, Lumbosacral
Keywords: lumbosacral radicular pain; pulsed radiofrequency; Alpha Lipoic acid
MeSH Terms: interventions — Pulsed Radiofrequency Treatment; Thioctic Acid; Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): Each patient in this group was treated with pulsed radiofrequency on the affected dorsal root ganglion at 42°C for 120 seconds
  Interventions: Procedure: pulsed radiofrequency
- Group II (Active Comparator): Each patient in this group was treated with pulsed radiofrequency as in group I plus oral alpha lipoic acid (ALA) 600 mg.
  Interventions: Drug: pulsed radiofrequency plus alpha lipoic acid

INTERVENTIONS:
Procedure: pulsed radiofrequency — Each patient in this group was treated with PRFT on the affected DRG at 42°C for 120 seconds.
  Other Names: PRF
  Arms: Group I
Drug: pulsed radiofrequency plus alpha lipoic acid — Each patient in this group was treated with PRFT as in group I plus oral alpha lipoic acid (ALA) 600 mg (Thiotacid 600 mg, EVA PHARMA, Egypt) three times per day (1800mg/day) for 3 weeks then 600mg once daily for 2 weeks.
  Other Names: PRF + ALA
  Arms: Group II

SUMMARY:
In this study, we try to evaluate the effect of using ALA as an adjuvant treatment in patients scheduled for pulsed radiofrequency treatment (PRFT) of the affected dorsal root ganglion (DRG) for treatment of Lumbo-Sacral radicular pain.

DETAILED DESCRIPTION:
Study design: The study is prospective, randomized, and open label started in August 2013 and was completed in March 2017 at Assiut University Hospital, Pain Unit after local ethical committee approval. All patients were informed verbally and in writing about the study, and they signed a detailed written informed consent about the procedure and the nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with severe chronic lumbo-sacral radicular pain of more than 6 months duration, not responding to medical treatment, and their Pain scores were > 7 were included in the study.

Exclusion Criteria:

* coagulopathy, surgical interference, advanced malignancy, known concurrent neurological or neurodegenerative disease, including those with impaired neurotransmission e.g. myasthenia gravis, multiple sclerosis, spinal cord injury, breastfeeding or pregnancy, allergy/sensitivity to lidocaine anesthetic or/ and non-ionic contrast media or/and steroid therapy, active psychiatric or mental conditions and uncontrolled medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NRS) | Before treatment
  The pain was evaluated using standard 10-point Numerical Pain Rating Scale (NRS) with 0 being no pain, and 10 representing the worst pain imaginable.
Numerical Pain Rating Scale (NRS) | 3 months after treatment
  The pain was evaluated using standard 10-point Numerical Pain Rating Scale (NRS) with 0 being no pain, and 10 representing the worst pain imaginable.
Numerical Pain Rating Scale (NRS) | 6 months after treatment
  The pain was evaluated using standard 10-point Numerical Pain Rating Scale (NRS) with 0 being no pain, and 10 representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, M.D., Principal Investigator — Assiut University faculty of medicine
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Boxem K, Cheng J, Patijn J, van Kleef M, Lataster A, Mekhail N, Van Zundert J. 11. Lumbosacral radicular pain. Pain Pract. 2010 Jul-Aug;10(4):339-58. doi: 10.1111/j.1533-2500.2010.00370.x. Epub 2010 May 17. PMID 20492580